CLINICAL TRIAL: NCT06863818
Title: Overcoming Resistance to EGFR Neutralization by Combination of Monoclonal Antibodies and Novel Cancer Drugs (Superamento Della Resistenza Alla Neutralizzazione di EGFR Nel Trattamento Con Anticorpi Monoclonali e Nuovi Farmaci Oncologici)
Brief Title: Overcoming Resistance to EGFR Neutralization by Combination of Monoclonal Antibodies and Novel Cancer Drugs
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: OROLCT; RC-2022-2773347 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2025-01-10; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: EGFR mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma and tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is aimed at patients with advanced cancer and EGFR mutation. Some molecules recently discovered at the level of tumor tissue can influence the response to anti-EGFR drugs. Among these molecules is NRG1, which binds to the EGFR receptor family.

Unravelling the mechanisms that give cancer cells resistance to such biologics could improve response to therapy and survival. And analyzing tumors during anti-EGFR drug therapy used in clinical practice could allow us to perform analyses on NRG1 and hypothesize a possible strategy to increase survival

DETAILED DESCRIPTION:
Experimental, tissue study. Patients with EGFR receptor amplification/overexpression or activating mutations treated with anti-EGFR cancer therapies will be involved in the study as required in normal clinical practice. Clinical information of the patients, relevant to the conduct of the study, will be collected: age, sex, ethnicity, smoking habit, diagnosis, staging of the tumor, site of any metastases, possible presence of ascites and/or pleural effusion, type of oncological therapy administered, concomitant therapies, radiological re-evaluation of the tumor, response to treatment, survival.

Similarly, peripheral blood, tissue obtained from archival tumor biopsies, ascitic and/or pleural fluid samples (taken, if present, as per clinical practice) will be collected. Primary cell cultures will be derived from tumor biopsies, ascites, and/or pleural effusion for in vitro studies The lymphocyte population will be isolated from the peripheral blood of patients

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥ 18 years
* patients with advanced cancer characterized by amplification/overexpression or activating mutations of the EGFR receptor.
* patients who are candidates for treatment with TKI and/or mAbs both in the first and second line, according to clinical practice.
* possibility of obtaining all information relating to the clinical history - obtaining written informed consent

Exclusion Criteria:

* Patients who in the opinion of the investigator may not be compliant with the needs of the study
* patients suffering from pathologies (e.g. psychiatric, neurological) that do not allow the obtaining of valid informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have EGFR receptor amplification/overexpression or activating mutations, either responsive to anti-EGFR therapy (TKIs or mABs) or recurrent despite anti-EGFR therapy (TKIs or mABs), will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate in vitro the molecular mechanisms that regulate the expression of NRG1 and/or IL-1 in relation to ERBB family receptors (EGFR, HER2, HER3 and HER4) before and after the standard therapy resistance phase in patients with mutation in | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  The expression of NRG1 and receptors of the ERBB family, pre- and post-treatment, and any receptors involved in resistance, including c-MET, IL-1R1, IL-1 and PD-L1, will be evaluated on tumor tissue. A qualitative and quantitative comparative evaluation of the expression of these genes between T0 and T2 will then be carried out.
  The expression of some cytokines including IL-1 and NRG1, at the T0, T1 and T2 timepoints, will be assessed by ELISA on blood and effusions (ascites, pleural fluid).

SECONDARY OUTCOMES:
To evaluate the response to TKIs and/or mAbs of isolated tumor tissue before and after the resistance phase to standard therapy in patients with EGFR mutation and propagated in vitro, in the presence of the lymphocyte component (T lymphocytes). The devel | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  To evaluate how the different isolated T population, before and after the onset of resistance, is able to influence the efficacy of therapies tested in vitro. We will use a 1:10 ratio of cancer cells to T lymphocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ardizzoni, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No